CLINICAL TRIAL: NCT06428136
Title: Comparative Effects of Clamshell Technique With Electrical Muscle Stimulation Versus Conservative Treatment in Iliotibial Band Tightness for Pain and Function
Brief Title: Comparative Effects of Clamshell Technique With EMS vs CTin Iliotibial Band Tightness for Pain and Function
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/709
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Tibial Muscular Dystrophy
MeSH Terms: conditions — Distal Myopathies | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clamshell exercises with Electrical Muscle Stimulation (CT + EMS) (Experimental)
  Interventions: Diagnostic Test: Clamshell exercises with Electrical Muscle Stimulation (CT + EMS)
- Conservative Treatment (CT) (Other)
  Interventions: Other: Conservative Treatment (CT)

INTERVENTIONS:
Diagnostic Test: Clamshell exercises with Electrical Muscle Stimulation (CT + EMS) — Side-lying clamshells: 3 sets of 10 repetitions per leg, 3 times per week Hip abduction with theraband: 3 sets of 10 repetitions per leg, 3 times per week Bridge with hip abduction: 3 sets of 10 repetitions per leg, 3 times per week
  Electrical muscle stimulation:
  Applied to the gluteus medius and minimus muscles for 20 minutes per session, 3 times per week Frequency and intensity adjusted to individual tolerance
  Arms: Clamshell exercises with Electrical Muscle Stimulation (CT + EMS)
Other: Conservative Treatment (CT) — Stretching: Iliotibial band stretch: 30-second hold, 3 repetitions per leg, 2 times per day Quadriceps stretch: 30-second hold, 3 repetitions per leg, 2 times per day Hamstring stretch: 30-second hold, 3 repetitions per leg, 2 times per day
  Arms: Conservative Treatment (CT)

SUMMARY:
Iliotibial band syndrome (ITBS) is a common knee injury that usually presents with pain and/or tenderness on palpation of the lateral aspect of the knee, superior to the joint line and inferior to the lateral femoral epicondyle. The current theory is that this condition is likely to be caused by compression of the innervated tissues beneath the iliotibial band (ITB), leading to inflammation.

DETAILED DESCRIPTION:
There were effects of clamshell exercises on gluteus medius, quadratus lumborum and anterior hip flexor. However their effect was limited on iliotibial band tightness. Hip/knee coordination and running style have also been identified as key factors in the treatment of ITBS, highlighting the complexity of the condition. The present study will focus on effect of clamshell techniques with electrical muscle stimulation versus Conservative treatment in iliotibial band tightness for pain and function.The goal is to determine which technique is more effecient in improving function and reducing pain and soreness of Iliotibial band.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45-65 years old (Jeong et al., 2019)
* Both genders will be included (Jeong et al., 2019)
* Diagnosed with iliotibial band tightness (ITBT) based on clinical examination and positive Noble compression test (Hutchinson et al., 2022)
* Reporting lateral knee pain aggravated by activity (Hutchinson et al., 2022)

Exclusion Criteria:

* Recent history of knee surgery or other knee injuries (Peterson et al., 2022)
* Presence of other musculoskeletal conditions affecting the knee (Peterson et al., 2022)
* Inflammatory conditions such as rheumatoid arthritis or gout (Peterson et al., 2022)
* Neurological conditions affecting leg function (Peterson et al., 2022)
* Pregnancy (Jeong et al., 2019)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Measured using a numeric pain rating scale (NPRS) | 12 Months
  ranging from 0 (no pain) to 10 (worst imaginable pain) assessed at baseline, after intervention, and at 1-month follow-up.
Lower Extremity Functional Scale (LEFS) | 12 months
  Measured using the Lower Extremity Functional Scale (LEFS) assessed at baseline, after intervention, and at 1-month follow-up
ITBT length | 12 months
  Measured using a goniometer at baseline, after intervention, and at 1-month follow-up.
Range of motion (ROM): | 12 months
  Measured using a goniometer for knee flexion and extension at baseline, after intervention, and at 1-month follow-up."

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No